CLINICAL TRIAL: NCT01425723
Title: An Open-Label, Multicenter, Evaluation of the Long-Term Safety and Efficacy of Recombinant Human Coagulation Factor IX Fusion Protein (rFIXFc) in the Prevention and Treatment of Bleeding Episodes in Previously Treated Subjects With Hemophilia B
Brief Title: Long-Term Safety and Efficacy of rFIXFc in the Prevention and Treatment of Bleeding Episodes in Previously Treated Participants With Hemophilia B
Acronym: B-YOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9HB01EXT; 2011-003075-11
Record Dates: First submitted 2011-08-19; First posted 2011-08-30 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2018-11

CONDITIONS: Severe Hemophilia B
Keywords: B-LONG; B-YOND; B-LONG Extension; rFIXFc; Severe Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — factor IX Fc fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- On-Demand (Experimental): The individual dose of rFIXFc to treat bleeding episodes will be based on participant's clinical condition, type and severity of the bleeding event, and if indicated, Factor IX peak (recovery) levels.
  Interventions: Biological: rFIXFc
- Prophylaxis (Experimental): Weekly prophylaxis, individualized prophylaxis or personalized prophylaxis available.
  Interventions: Biological: rFIXFc

INTERVENTIONS:
Biological: rFIXFc — Administered as specified in the treatment arm.
  Other Names: coagulation factor IX (recombinant) Fc fusion protein; Alprolix; BIIB029

SUMMARY:
The primary objective of the study is to evaluate the long-term safety of rFIXFc in participants with hemophilia B.

The secondary objective of this study is to evaluate the efficacy of rFIXFc in the prevention and treatment of bleeding episodes.

DETAILED DESCRIPTION:
Participants will follow either a prophylaxis or on-demand regimen. The starting dose in this study will be determined by the clinical profile of the patient in the preceding studies, B-LONG 998HB102 (NCT01027364) and Kids B-LONG study 9HB02PED (NCT01440946)

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects who have completed studies 998HB102 (NCT01027364) or 9HB02PED (NCT01440946) or other studies with rFIXFc
* Ability to understand the purposes & risks of the study and provide signed and dated informed consent.

Key Exclusion Criteria:

* High-titer inhibitor (>/=5.00 BU/mL)

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-12-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Bioverativ Therapeutics Inc.
Locations (49):
- United States (10):
  - Research Site, Phoenix, Arizona
  - Research Site, Sacramento, California
  - Research Site, Aurora, Colorado
  - Research Site, Atlanta, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Indianapolis, Indiana
  - Research Site, New Orleans, Louisiana
  - Research Site, East Lansing, Michigan
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Seattle, Washington
- Australia (4):
  - Research Site, Adelaide, South Australia
  - Research site, Parkville, Victoria
  - Research site, Murdoch, Western Australia
  - Research Site, Perth, Western Australia
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Leuven
- Research Site, Campinas, São Paulo, Brazil
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (4):
  - Research Site, Beijing, Beijingshì
  - Research Site, Guangzhou, Guangdongsheng
  - Research Site, Shanghai, Shànghaishì
  - Research Site, Tianjing, Tianjinshì
- Research Site, Marseille, Bouches-Du-Rhône, France
- Research Site, Bonn, North Rhine-Westphalia, Germany
- Hong Kong (2):
  - Research Site, Hong Kong, New Territories
  - Research site, Hong Kong
- India (3):
  - Research Site, Bangalore, Karnataka
  - Research Site, Pune, Maharashtra
  - Research Site, Vellore, Tamil Nadu
- Research Site, Dublin, Ireland
- Italy (2):
  - Research Site, Florence
  - Research Site, Milan
- Japan (6):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Kitakyushu, Fukuoka
  - Research Site, Kawasaki, Kanagawa
  - Research Site, Kashihara-shi, Nara
  - Research Site, Shinjuku-ku, Tokyo-To
  - Research Site, Tokyo, Tokyo-To
- Research Site, Utrecht, Netherlands
- Research Site, Lodz, Poland
- South Africa (2):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Cape Town, Western Cape
- Sweden (2):
  - Research Site, Malmo
  - Research Site, Stockholm
- United Kingdom (4):
  - Research Site, Cambridge, Cambridgeshire
  - Research Site, London, Greater London
  - Research site, London, Greater London
  - Research Site, Basingstoke, Hampshire

REFERENCES:
- [Derived] Astermark J, Hermans C, Ezzalfani M, Sidhom A, Barbier S, Kragh N, Falk A, Eriksson D. Recombinant factor IX Fc prophylaxis reduces pain and increases levels of physical activity, with sustained, long-term improvements in patients with hemophilia B: post hoc analysis of phase III trials using patient-reported outcomes. Ther Adv Hematol. 2023 May 29;14:20406207231170701. doi: 10.1177/20406207231170701. eCollection 2023. PMID 37283819
- [Derived] Shapiro AD, Kulkarni R, Ragni MV, Chambost H, Mahlangu J, Oldenburg J, Nolan B, Ozelo MC, Foster MC, Willemze A, Barnowski C, Jain N, Winding B, Dumont J, Lethagen S, Barnes C, Pasi KJ. Post hoc longitudinal assessment of the efficacy and safety of recombinant factor IX Fc fusion protein in hemophilia B. Blood Adv. 2023 Jul 11;7(13):3049-3057. doi: 10.1182/bloodadvances.2022009230. PMID 36848635
- [Derived] Shapiro AD, Pasi KJ, Ozelo MC, Kulkarni R, Barnowski C, Winding B, Szamosi J, Lethagen S. Extending recombinant factor IX Fc fusion protein dosing interval to 14 or more days in patients with hemophilia B. Res Pract Thromb Haemost. 2018 Nov 29;3(1):109-113. doi: 10.1002/rth2.12163. eCollection 2019 Jan. PMID 30656283

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed either of the Phase 3 studies (Study 998HB102 [NCT01027364], Study 9HB02PED [NCT01440946]) were expected to be eligible to enroll in this study.
Groups:
- rFIXFc (Participants From 9HB02PED): Participants received Recombinant Human Coagulation Factor IX Fusion Protein (rFIXFc) intravenously (IV) according to their assigned treatment regimen as follows: Weekly prophylaxis (P): Participants received 20 IU/kg to 100 IU/kg rFIXFc once weekly. Dose was based on participants clinical profile in parent study and individual pharmacokinetic profile, trough and/or peak (recovery) values; Individualized P: 100 IU/kg rFIXFc every 8 to 16 days or twice a month; Personalized P: included addition of prevention doses prior to strenuous activity; targeting FIX trough level of greater than (>)5%, if warranted by bleeding history and/or activity level or dosing twice a week (25 IU/kg twice weekly versus 50 IU/kg once weekly) for participants who may have better control with such regimen. Participants who reached age of 12 during study could also choose to switch to episodic treatment group, with dosing based on participants clinical condition and type and severity of bleeding event.
- rFIXFc (Participants From 998HB102): Participants received rFIXFc IV according to their assigned treatment regimen as follows: Weekly prophylaxis: Participants received 20 international units per kilogram (IU/kg) to 100 IU/kg rFIXFc once weekly. Dose was based on participants clinical profile observed in parent study and individual pharmacokinetic profile, trough, and/or peak (recovery) values. Individualized prophylaxis: 100 IU/kg rFIXFc every 8 to 16 days or twice a month; Personalized Prophylaxis: included addition of prevention doses prior to strenuous activity; targeting a FIX trough level of > 5 percent (%), if warranted by the bleeding history and/or activity level or dosing twice a week (25 IU/kg, twice weekly, versus 50 IU/kg, once weekly) for participants who may have better control with such a regimen. Episodic (On Demand): The individual dose of rFIXFc to treat bleeding episodes was based on participants clinical condition, type and severity of the bleeding event.
Period: Overall Study
Arm/Group | rFIXFc (Participants From 9HB02PED) | rFIXFc (Participants From 998HB102)
Started | 27 (13 participants in <6 Years Old Age Cohort and 14 participants in 6 to <12 Years Old Age Cohort.) | 93
Weekly Prophylaxis | 23 | 51
Individualized Prophylaxis | 5 | 31
Personalized Prophylaxis | 2 | 17
Episodic | 0 | 15
Surgery Subgroup (Participants who have undergone major surgery or have major surgical/rehabilitation period in study.) | 1 | 15
Completed | 23 | 75
Not Completed | 4 | 18
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 0 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Other | 1 | 10

BASELINE CHARACTERISTICS:
Groups:
- rFIXFc (Participants From 9HB02PED): Participants received rFIXFc IV according to their assigned treatment regimen as follows: Weekly prophylaxis (P): Participants received 20 IU/kg to 100 IU/kg rFIXFc once weekly. Dose was based on participants clinical profile in parent study and individual pharmacokinetic profile, trough and/or peak (recovery) values; Individualized P: 100 IU/kg rFIXFc every 8 to 16 days or twice a month; Personalized P: included addition of prevention doses prior to strenuous activity; targeting FIX trough level of >5%, if warranted by bleeding history and/or activity level or dosing twice a week (25 IU/kg twice weekly versus 50 IU/kg once weekly) for participants who may have better control with such regimen. Participants who reached age of 12 during study could also choose to switch to episodic treatment group, with dosing based on participants clinical condition and type and severity of bleeding event.
- rFIXFc (Participants From 998HB102): Participants received rFIXFc IV according to their assigned treatment regimen as follows: Weekly prophylaxis: Participants received 20 IU/kg to 100 IU/kg rFIXFc once weekly. Dose was based on participants clinical profile observed in parent study and individual pharmacokinetic profile, trough, and/or peak (recovery) values. Individualized prophylaxis: 100 IU/kg rFIXFc every 8 to 16 days or twice a month; Personalized Prophylaxis: included addition of prevention doses prior to strenuous activity; targeting a FIX trough level of > 5%, if warranted by the bleeding history and/or activity level or dosing twice a week (25 IU/kg, twice weekly, versus 50 IU/kg, once weekly) for participants who may have better control with such a regimen. Episodic (On Demand): The individual dose of rFIXFc to treat bleeding episodes was based on participants clinical condition, type and severity of the bleeding event.
- Total: Total of all reporting groups
Arm/Group | rFIXFc (Participants From 9HB02PED) | rFIXFc (Participants From 998HB102) | Total
Number analyzed (Participants) | 27 | 93 | 120
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 27 | 8 | 35
  Between 18 and 65 years | 0 | 85 | 85
  > 65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 27 | 93 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 11 | 11
  Not Hispanic or Latino | 27 | 78 | 105
  Unknown or Not Reported | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19 | 47 | 66
  Black or African American | 2 | 9 | 11
  Asian | 5 | 27 | 32
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Other | 1 | 10 | 11
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Positive Inhibitor Development
Description: An inhibitor test result greater than or equal to (>=)0.6 Bethesda units per milliliter (BU/mL), confirmed on 2 separate samples drawn 2 to 4 weeks apart, was considered positive. Both tests were to be performed by the central laboratory using the Nijmegen-modified Bethesda Assay. Data was summarized by treatment regimen for participants from Study 998HB102 and by age cohort (<6 years and 6 to <12 years old) and treatment regimen for participants from Study 9HB02PED per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Approximately 5 years
Population: Safety Analysis Set included participants who received at least 1 dose of Recombinant Human Coagulation Factor IX Fusion Protein (rFIXFc) in study 9HB01EXT.
Measure: Count of Participants; unit: Participants
Groups:
- rFIXFc (9HB02PED [<6 Years Old]): Participants with less than (<) 6 years old age received rFIXFc IV according to their assigned treatment regimen as follows: Weekly prophylaxis (P): 20 IU/kg to 100 IU/kg rFIXFc once weekly. Dose was based on participants clinical profile in parent study and individual pharmacokinetic profile, trough and/or peak (recovery) values; Individualized P: 100 IU/kg rFIXFc every 8 to 16 days or twice a month; Personalized P: included addition of prevention doses prior to strenuous activity; targeting FIX trough level of > 5%, if warranted by bleeding history and/or activity level or dosing twice a week (25 IU/kg, twice weekly, versus 50 IU/kg, once weekly) for participants who may have better control with such a regimen. Participants who reached age of 12 during study could also choose to switch to episodic treatment group, with dosing based on participants clinical condition and type and severity of bleeding event.
- rFIXFc (9HB02PED [6 to <12 Years]): Participants with 6 to <12 years old age received rFIXFc IV according to their assigned treatment regimen as follows: Weekly prophylaxis (P): 20 IU/kg to 100 IU/kg rFIXFc once weekly. Dose was based on participants clinical profile in parent study and individual pharmacokinetic profile, trough and/or peak (recovery) values; Individualized P: 100 IU/kg rFIXFc every 8 to 16 days or twice a month; Personalized P: included addition of prevention doses prior to strenuous activity; targeting FIX trough level of > 5%, if warranted by bleeding history and/or activity level or dosing twice a week (25 IU/kg, twice weekly, versus 50 IU/kg, once weekly) for participants who may have better control with such regimen. Participants who reached age of 12 during study could also choose to switch to episodic treatment group, with dosing based on participants clinical condition and type and severity of bleeding event.
Arm/Group | rFIXFc (9HB02PED [<6 Years Old]) | rFIXFc (9HB02PED [6 to <12 Years]) | rFIXFc (Participants From 998HB102)
Number analyzed (Participants) | 13 | 14 | 93
Participants | 0 | 0 | 0

2. Secondary Outcome: Annualized Bleeding Rate (ABR)
Description: ABR is annualized number of bleeding episodes per participant per year. Bleeding episodes were classified as spontaneous if participant records bleeding event when there is no known contributing factor such as definite trauma/antecedent strenuous activity and classified as traumatic if participant records bleeding event when there is known reason for bleed. ABR=(Number of bleeding episodes during efficacy period/number of days during efficacy period)*365.25. Efficacy period reflects sum of all intervals of time during which participants were treated with rFIXFc per treatment regimen excluding major and minor surgical/rehabilitation periods and large injection intervals. ABR was summarized by treatment regimen for participants from study 998HB102 and by age cohort (<6 years and 6 to <12 years old) and treatment regimen for participants from study 9HB02PED per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Approximately 5 years
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of rFIXFc. Here 'n' (number analyzed) signifies number of participants who were analyzed in each treatment regimen, for each arm, respectively.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Groups:
- rFIXFc (9HB02PED [<6 Years Old Age Cohort]): Participants with < 6 years old age received rFIXFc IV according to their assigned treatment regimen as follows: Weekly prophylaxis (P): 20 IU/kg to 100 IU/kg rFIXFc once weekly. Dose was based on participants clinical profile in parent study and individual pharmacokinetic profile, trough and/or peak (recovery) values; Individualized P: 100 IU/kg rFIXFc every 8 to 16 days or twice a month; Personalized P: included addition of prevention doses prior to strenuous activity; targeting FIX trough level of > 5%, if warranted by bleeding history and/or activity level or dosing twice a week (25 IU/kg, twice weekly, versus 50 IU/kg, once weekly) for participants who may have better control with such a regimen. Participants who reached age of 12 during study could also choose to switch to episodic treatment group, with dosing based on participants clinical condition and type and severity of bleeding event.
- rFIXFc (9HB02PED [6 to <12 Years Old Age Cohort]): Participants with 6 to <12 years old age received rFIXFc IV according to their assigned treatment regimen as follows: Weekly prophylaxis (P): 20 IU/kg to 100 IU/kg rFIXFc once weekly. Dose was based on participants clinical profile in parent study and individual pharmacokinetic profile, trough and/or peak (recovery) values; Individualized P: 100 IU/kg rFIXFc every 8 to 16 days or twice a month; Personalized P: included addition of prevention doses prior to strenuous activity; targeting FIX trough level of > 5%, if warranted by bleeding history and/or activity level or dosing twice a week (25 IU/kg, twice weekly, versus 50 IU/kg, once weekly) for participants who may have better control with such regimen. Participants who reached age of 12 during study could also choose to switch to episodic treatment group, with dosing based on participants clinical condition and type and severity of bleeding event.
- rFIXFc (Participants From Study 998HB102): Participants received rFIXFc IV according to their assigned treatment regimen as follows: Weekly prophylaxis: Participants received 20 IU/kg to 100 IU/kg rFIXFc once weekly. Dose was based on participants clinical profile observed in parent study and individual pharmacokinetic profile, trough, and/or peak (recovery) values. Individualized prophylaxis: 100 IU/kg rFIXFc every 8 to 16 days or twice a month; Personalized Prophylaxis: included addition of prevention doses prior to strenuous activity; targeting a FIX trough level of > 5%, if warranted by the bleeding history and/or activity level or dosing twice a week (25 IU/kg, twice weekly, versus 50 IU/kg, once weekly) for participants who may have better control with such a regimen. Episodic (On Demand): The individual dose of rFIXFc to treat bleeding episodes was based on participants clinical condition, type and severity of the bleeding event.
Arm/Group | rFIXFc (9HB02PED [<6 Years Old Age Cohort]) | rFIXFc (9HB02PED [6 to <12 Years Old Age Cohort]) | rFIXFc (Participants From Study 998HB102)
Number analyzed (Participants) | 13 | 14 | 93
episodes per participant per year
  Weekly Prophylaxis: number analyzed (Participants) | 13 | 10 | 51
  Weekly Prophylaxis | 1.04 [0.00 to 2.28] | 1.14 [0.54 to 2.34] | 2.26 [0.40 to 5.16]
  Individualized Prophylaxis: number analyzed (Participants) | 0 | 5 | 31
  Individualized Prophylaxis |  | 3.69 [3.54 to 5.21] | 1.85 [0.76 to 4.00]
  Personalized Prophylaxis: number analyzed (Participants) | 1 | 1 | 16
  Personalized Prophylaxis | 0.54 [0.54 to 0.54] | 3.13 [3.13 to 3.13] | 2.91 [1.14 to 5.36]
  Episodic: number analyzed (Participants) | 0 | 0 | 15
  Episodic |  |  | 11.64 [5.12 to 18.54]

3. Secondary Outcome: Annualized Spontaneous Joint Bleeding Episodes
Description: Bleeding episodes were classified as spontaneous if participant records a bleeding event when there is no known contributing factor such as definite trauma/antecedent strenuous activity. In addition, location of bleed (joint, internal, skin/mucosa or muscle) were also collected. Annualized spontaneous joint bleeding episodes=(Number of spontaneous joint bleeding episodes during efficacy period/number of days during efficacy period)*365.25. Efficacy period reflects sum of all intervals of time during which participants were treated with rFIXFc per treatment regimen excluding major and minor surgical/rehabilitation periods and large injection intervals. Bleeding episodes were summarized by treatment regimen for participants from study 998HB102 and by age cohort (<6 years and 6 to <12 years old) and treatment regimen for participants from study 9HB02PED as per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Approximately 5 years
Population: FAS included all participants who received at least 1 dose of rFIXFc. Here 'n' (number analyzed) signifies number of participants who were analyzed in each treatment regimen, for each arm, respectively.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | rFIXFc (9HB02PED [<6 Years Old Age Cohort]) | rFIXFc (9HB02PED [6 to <12 Years Old Age Cohort]) | rFIXFc (Participants From Study 998HB102)
Number analyzed (Participants) | 13 | 14 | 93
episodes per participant per year
  Weekly Prophylaxis: number analyzed (Participants) | 13 | 10 | 51
  Weekly Prophylaxis | 0.00 [0.00 to 1.06] | 0.00 [0.00 to 1.40] | 0.38 [0.00 to 2.25]
  Individualized Prophylaxis: number analyzed (Participants) | 0 | 5 | 31
  Individualized Prophylaxis |  | 0.00 [0.00 to 0.29] | 0.38 [0.00 to 1.43]
  Personalized Prophylaxis: number analyzed (Participants) | 1 | 1 | 16
  Personalized Prophylaxis | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.30 [0.00 to 1.37]
  Episodic: number analyzed (Participants) | 0 | 0 | 15
  Episodic |  |  | 2.15 [0.58 to 11.68]

4. Secondary Outcome: Total Number of Exposure Days (EDs)
Description: An exposure day is a 24-hour period in which one or more rFIXFc injections are given. The total number of days of exposure to rFIXFc were summarized by treatment regimen for participants from study 998HB102 and by age cohort (<6 years and 6 to <12 years old) and treatment regimen for participants from study 9HB02PED as per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Approximately 5 years
Population: Safety Analysis Set included participants who received at least 1 dose of rFIXFc in study 9HB01EXT. Here 'n' (number analyzed) signifies number of participants who were analyzed in each treatment regimen, for each arm, respectively.
Measure: Median (Full Range); unit: days
Arm/Group | rFIXFc (9HB02PED [<6 Years Old Age Cohort]) | rFIXFc (9HB02PED [6 to <12 Years Old Age Cohort]) | rFIXFc (Participants From Study 998HB102)
Number analyzed (Participants) | 13 | 14 | 93
days
  Weekly Prophylaxis: number analyzed (Participants) | 13 | 10 | 51
  Weekly Prophylaxis | 55.00 [8.0 to 176.0] | 165.00 [3.0 to 202.0] | 169.00 [4.0 to 327.0]
  Individualized Prophylaxis: number analyzed (Participants) | 0 | 5 | 31
  Individualized Prophylaxis |  | 54.00 [4.0 to 141.0] | 110.00 [9.0 to 369.0]
  Personalized Prophylaxis: number analyzed (Participants) | 1 | 1 | 17
  Personalized Prophylaxis | 157.00 [157.00 to 157.00] | 90.00 [90.00 to 90.00] | 146.00 [7.0 to 431.0]
  Episodic: number analyzed (Participants) | 0 | 0 | 15
  Episodic |  |  | 52.00 [0.0 to 164.0]

5. Secondary Outcome: Annualized rFIXFc Consumption (International Units Per Kilogram [IU/kg])
Description: Annualized consumption = (total international unit per kilogram [IU/kg] of study treatment received during the efficacy period / total number of days during the efficacy period) multiplied by 365.25. Efficacy period reflects sum of all intervals of time during which participants were treated with rFIXFc per treatment regimen excluding major and minor surgical/rehabilitation periods and large injection intervals. Annualized consumption was summarized by treatment regimen for participants from study 998HB102 and by age cohort (<6 years and 6 to <12 years old) and treatment regimen for participants from study 9HB02PED as per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Approximately 5 years
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: IU per kilogram per participant per year
Arm/Group | rFIXFc (9HB02PED [<6 Years Old Age Cohort]) | rFIXFc (9HB02PED [6 to <12 Years Old Age Cohort]) | rFIXFc (Participants From Study 998HB102)
Number analyzed (Participants) | 13 | 14 | 93
IU per kilogram per participant per year
  Weekly Prophylaxis: number analyzed (Participants) | 13 | 10 | 51
  Weekly Prophylaxis | 3382.5 [2930.9 to 3667.4] | 3212.0 [2838.5 to 3344.4] | 2598.0 [2129.8 to 3370.9]
  Individualized Prophylaxis: number analyzed (Participants) | 0 | 5 | 31
  Individualized Prophylaxis |  | 3700.7 [3689.2 to 3716.5] | 2894.8 [2520.0 to 4023.5]
  Personalized Prophylaxis: number analyzed (Participants) | 1 | 1 | 16
  Personalized Prophylaxis | 3331.7 [3331.7 to 3331.7] | 8931.2 [8931.2 to 8931.2] | 3671.2 [2394.8 to 5563.3]
  Episodic: number analyzed (Participants) | 0 | 0 | 15
  Episodic |  |  | 595.6 [363.8 to 1024.5]

6. Secondary Outcome: Physicians' Global Assessment of Participant's Response to rFIXFc Regimen Using a 4-Point Scale
Description: Participants were assessed for response to their rFIXFc regimen using following 4-point scale: 1=Excellent: bleeding episodes responded to less than or equal to (<=)usual number of injections or dose of rFIXFc or rate of breakthrough bleeding during prophylaxis was <= that usually observed; 2=Effective: most bleeding episodes responded to same number of injections and dose, but some required more injections or higher doses, or there was minor increase in rate of breakthrough; 3=Partially Effective: bleeding episodes most often required more injections and/or higher doses than expected or adequate breakthrough bleeding prevention during prophylaxis required more frequent injections and/or higher doses and 4=Ineffective: routine failure to control hemostasis/hemostatic control require additional agents. Total number of scale responses =total count of scale responses for all participants; multiple responses per participant including those at scheduled and unscheduled visits are counted.
Time Frame: Approximately 5 years
Population: FAS included all participants who received at least 1 dose of rFIXFc. Data was summarized by treatment regimen for participants from Study 998HB102 and Study 9HB02PED per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Measure: Count of Units; unit: Responses
Units Other Than Participants: Responses
Arm/Group | rFIXFc (Participants From 9HB02PED) | rFIXFc (Participants From 998HB102)
Number analyzed (Participants) | 27 | 93
Number analyzed (Responses) | 151 | 815
Responses
  Excellent | 131 | 622
  Effective | 19 | 184
  Partially Effective | 1 | 9
  Ineffective | 0 | 0

7. Secondary Outcome: Participant's Assessment of Response (Excellent or Good Response) to rFIXFc Injections for the Treatment of Bleeding Episodes Using a 4-Point Scale
Description: Using eDiary, participant received rating for treatment response to any bleeding episode (BE) using 4-point scale- 1=Excellent: Abrupt pain relief and/or improvement in signs of bleeding within approximately (approx.) 8 hours (h) after initial injection (inj.); 2=Good: Definite pain relief and/or improvement in signs of bleeding within approx. 8h after an injection, but possibly requiring more than 1 injection after 24-48h for complete resolution; 3=Moderate: Probable/slight beneficial effect within 8h after initial injection and requires more than 1 injection and 4=None: No improvement, or condition worsens within approx. 8h after initial injection. This assessment was to be made approx. 8 to 12h from time the injection was given to treat BE and prior to any additional doses of rFIXFc given for same bleeding episode. Percentages are based on the number of bleeding episodes for which a response (excellent or good) was provided for the first injection during the efficacy period.
Time Frame: Approximately 5 years
Population: FAS was analyzed. Data was summarized by treatment regimen for participants from study 998HB102 and by age cohort (<6 years and 6 to <12 years old) and treatment regimen for participants from study 9HB02PED per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Measure: Count of Units; unit: Injections
Units Other Than Participants: Injections
Arm/Group | rFIXFc (9HB02PED [<6 Years Old Age Cohort]) | rFIXFc (9HB02PED [6 to <12 Years Old Age Cohort]) | rFIXFc (Participants From 998HB102)
Number analyzed (Participants) | 13 | 14 | 93
Number analyzed (Injections) | 75 | 90 | 1646
Injections
  Weekly Prophylaxis: number analyzed (Injections) | 74 | 57 | 461
  Weekly Prophylaxis | 60 | 47 | 342
  Individualized Prophylaxis: number analyzed (Injections) | 0 | 31 | 386
  Individualized Prophylaxis |  | 25 | 336
  Personalized Prophylaxis: number analyzed (Injections) | 1 | 2 | 178
  Personalized Prophylaxis | 0 | 1 | 135
  Episodic: number analyzed (Injections) | 0 | 0 | 621
  Episodic |  |  | 603

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent Form (ICF) through follow-up (approximately 5 years)
Description: Adverse events (AEs) data was planned to be reported for each group and for the overall participants. AEs emergent during major surgical/rehabilitation periods are analyzed separately as per planned analysis and are presented as separate groups.
Groups:
- Overall rFIXFc (Participants From 9HB02PED and 998HB102): All participants who received rFIXFc drug in study 9HB01EXT, from studies 9HB02PED and 998HB102 (combined). AEs emergent during major surgical/rehabilitation periods are excluded and are presented as separate groups.
- rFIXFc (Participants From 9HB02PED in Surgery Subgroup); rFIXFc (Participants From 998HB102 in Surgery Subgroup): Participants who required emergent or elective surgery while participating in this study and treated with the dose and regimen of rFIXFc as appropriate for the type of surgery. Participants returned to a regular rFIXFc regimen once all dosing for the postoperative rehabilitation period had been completed.
Arm/Group | rFIXFc (Participants From 9HB02PED) | rFIXFc (Participants From 998HB102) | Overall rFIXFc (Participants From 9HB02PED and 998HB102) | rFIXFc (Participants From 9HB02PED in Surgery Subgroup) | rFIXFc (Participants From 998HB102 in Surgery Subgroup)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/93 | 0/120 | 0/1 | 0/15
Serious Adverse Events (participants affected / at risk) | 5/27 | 31/93 | 36/120 | 0/1 | 1/15
Other Adverse Events (participants affected / at risk) | 23/27 | 66/93 | 89/120 | 0/1 | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rFIXFc (Participants From 9HB02PED) (N=27) | rFIXFc (Participants From 998HB102) (N=93) | Overall rFIXFc (Participants From 9HB02PED and 998HB102) (N=120) | rFIXFc (Participants From 9HB02PED in Surgery Subgroup) (N=1) | rFIXFc (Participants From 998HB102 in Surgery Subgroup) (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Necrotising retinitis (Eye disorders) | 0 | 1 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 3 | 3 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 4 | 7 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Slipping rib syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Posterior interosseous syndrome (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 2 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 2 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Victim of crime (Social circumstances) | 0 | 1 | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Anal Sphincter Atony (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rFIXFc (Participants From 9HB02PED) (N=27) | rFIXFc (Participants From 998HB102) (N=93) | Overall rFIXFc (Participants From 9HB02PED and 998HB102) (N=120) | rFIXFc (Participants From 9HB02PED in Surgery Subgroup) (N=1) | rFIXFc (Participants From 998HB102 in Surgery Subgroup) (N=15)
Hypertension (Vascular disorders) | 0 | 7 | 7 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 4 | 11 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 2 | 4 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 2 | 2 | 4 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 4 | 6 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 3 | 5 | 8 | 0 | 0
Serum ferritin decreased (Investigations) | 2 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 8 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 5 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 5 | 0 | 0
Seasonal allergy (Immune system disorders) | 4 | 3 | 7 | 0 | 0
Headache (Nervous system disorders) | 3 | 15 | 18 | 0 | 0
Pyrexia (General disorders) | 6 | 5 | 11 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 6 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 7 | 8 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 5 | 5 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 5 | 5 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 7 | 12 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 5 | 5 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 5 | 5 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 10 | 14 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0 | 0
Ear infection (Infections and infestations) | 3 | 1 | 4 | 0 | 0
Influenza (Infections and infestations) | 1 | 8 | 9 | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 5 | 5 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 1 | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 14 | 17 | 0 | 0
Paronychia (Infections and infestations) | 2 | 0 | 2 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 5 | 6 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 6 | 8 | 0 | 0
Varicella (Infections and infestations) | 2 | 1 | 3 | 0 | 0
Viral infection (Infections and infestations) | 2 | 3 | 5 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2013-11-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT01425723/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT01425723/SAP_001.pdf